CLINICAL TRIAL: NCT00999557
Title: Efficacy of Topical Bimatoprost in Promoting Hair Growth in the Region of the Eyebrow and Eyelashes for Post-chemotherapy Patients Versus Normal Patients
Brief Title: Bimatoprost Ophthalmic Solution in Increasing Eyebrow and Eyelash Growth in Patients Who Have Undergone Chemotherapy for Breast Cancer and in Healthy Participants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CDR0000657044; UCLA-0904044
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2016-04

CONDITIONS: Alopecia; Breast Cancer
Keywords: breast cancer; male breast cancer; alopecia
MeSH Terms: conditions — Alopecia; Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients apply topical bimatoprost ophthalmic solution to base of upper eyelid margins OR to eyebrow region once daily for 4 months in the absence of unacceptable toxicity.
  Interventions: Drug: bimatoprost ophthalmic solution
- Arm II (Placebo Comparator): Patients apply topical placebo solution to base of upper eyelid margins OR to eyebrow region once daily for 4 months in the absence of unacceptable toxicity.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution — Applied topically
  Arms: Arm I
Drug: placebo — Applied topically
  Arms: Arm II

SUMMARY:
RATIONALE: Bimatoprost ophthalmic solution may help increase eyebrow and eyelash growth in patients who have undergone chemotherapy.

PURPOSE: This randomized clinical trial is studying how wells bimatoprost ophthalmic solution works in increasing eyebrow and eyelash growth in patients who have undergone chemotherapy for breast cancer and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effectiveness of bimatoprost ophthalmic solution in expediting regrowth of eyebrows and eyelashes in patients who have undergone chemotherapy for breast cancer and in increasing eyebrow growth in healthy participants with no known underlying disease as assessed by two physicians and an aesthetics expert on a scale of 0-4.

Secondary

* To assess the effectiveness of this treatment as assessed by patient self-report on a scale of 0-4.
* To assess the psychological impact of this treatment as assessed by patient-completed questionnaires.

OUTLINE: Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients apply topical bimatoprost ophthalmic solution to base of upper eyelid margins OR to eyebrow region once daily for 4 months in the absence of unacceptable toxicity.
* Arm II: Patients apply topical placebo solution to base of upper eyelid margins OR to eyebrow region once daily for 4 months in the absence of unacceptable toxicity.

Patients complete questionnaires at baseline and monthly for 5 months about changes in eyebrows/eyelashes, side effects of treatment, and the psychological impact of treatment. Photographs of eyebrows or eyelashes and surrounding skin are taken at baseline and monthly for 5 months and reviewed by a physician and aesthetics expert.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Meets 1 of the following criteria:
* Diagnosis of breast cancer (group 1)
* Completed chemotherapy within the past month that has resulted in eyebrow alopecia or eyelash hypotrichosis
* Eyebrow score of 0-2 or eyelash score of 0-2 on the study's qualitative eyebrow or eyelash growth chart
* Has no known underlying disease (group 2)
* Desires thicker, fuller, or more numerous eyebrows

Exclusion criteria

* pregnant
* does not Speak a language adequately covered by study translator services
* cognitive impairment
* history of trauma or burn to the eyebrow region, alopecia areata, or trichotillomania
* known diagnoses possibly underlying or contributing to the state of the eyebrows including, but not limited to, telogen effluvium or anagen effluvium (group 2)
* active ocular disease (group 1)
* thyroid hormone level abnormalities (group 2)
* More than 2 years since prior ocular surgery (group 1)
* prior topical medication for increasing eyebrow growth within 30 days od starting study treatment
* concomitant chemotherapy for the treatment of cancer (group 1)
* concomitant therapy for eyelash or eyebrow growth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Measuring regrowth of eyebrows and eyelashes by Bimatoprost Opthalmic solution | every 30 days for 4 months
  Efficacy of Bimatoprost Opthalmic solution in expediting regrowth of eyebrows and eyelashes in patients who have undergone chemotherapy for breast cancer and in increasing eyebrow growth in healthy participants with no known underlying disease as assessed by two physicians and an aesthetics expert on a scale of 0-4.

SECONDARY OUTCOMES:
Effectiveness of Bimatoprost Ophthalmic Solution as assessed by patient self-report on a scale of 0-4. | every 30 days for 4 months
Psychological impact as assessed at baseline and at 6 months by patient-completed questionnaires | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Kim, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States